CLINICAL TRIAL: NCT04757051
Title: Real-life Use of BENART TM in Patients With Symptomatic Knee Osteoarthritis
Status: Completed | Type: Observational
Sponsor: TRB Chemedica AG (Industry)
Responsible Party: Sponsor
Other Study IDs: BEN-PMCF-DE-2020
Record Dates: First submitted 2021-02-11; First posted 2021-02-16 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2022-08

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
PMCF study to assess the effectiveness and safety of BENART in the treatment of symptomatic knee OA in a real-life clinical setting when used according to the instructions for use.

ELIGIBILITY:
Inclusion Criteria:

* male or female aged between 18 and 99 years
* diagnosis of symptomatic knee OA: Kellgren & Lawrence grade II/III
* physician's recommendation to use BENART TM prior to recruitment
* signed informed consent

Exclusion Criteria:

* known allergy or hypersensitivity to any of the BENART TM components
* infection or skin disease at or around the injection site
* severe Inflammation, synovitis, or arthritis of the knee joint and/or any other signs of inflammation (e.g. pain causing nocturnal awakenings, knee heat,...)
* history of autoimmune and crystal diseases (e.g. gout, pseudogout, hereditary hemochromatosis, ...)
* evidence of lymphatic or venous stasis or serious blood disorders
* known pregnancy or breast feeding
* significant joint effusion (confirmed by objective clinical signs and/or ultrasound and/or puncture)
* individuals who are unable to fully understand all aspects of the study that are relevant to the decision to participate, or who could be manipulated or unduly influenced as a result of a compromised position, expectation of benefits or fear of retaliatory response (including persons needing legally designated representatives, illiterate persons or persons with insufficient knowledge of local language)

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients between 18 and 99 years with knee osteoarthitis and a recommendation for treatment with BENART TM.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2021-03-11 (Actual); Primary Completion 2022-04-25 (Actual); Study Completion 2022-04-25 (Actual)

PRIMARY OUTCOMES:
Change of subjective therapy evaluation (KOOS questionnaire) compared to baseline | week 1, week 12, week 24, week 36
  Knee injury and Osteoarthritis Outcome Score (KOOS) to assess pain, other symptoms, activities of daily living (ADL), function in sport and recreation (Sport/Rec) and knee-related Quality of Life (QoL) on a 5-point Likert scale
Change of pain intensity compared to baseline (visual analogue scale, VAS) | week 1, week 12, week 24, week 36
  Evaluation of pain intensity by the patient on a 10 cm VAS-slider. 10 cm equals the worst pain.
Change of patient's global assessment (overall impression of clinical OA severity on a numerical rating scale from 0 to 10) | week 1, week 12, week 24, week 36
  The change of overall subjective symptom severity evaluation on a scale from 0 (very good condition) to 10 (very poor condition).
Change of clinical global impression (overall impression of clinical OA severity of the investigator on a numerical rating scale from 0 to 10) | week 1, week 12, week 24, week 36
  The change of clinical global Impression on a scale from 0 (very good condition) to 10 (very poor condition).
Responder rate according to OMERACT-OARSI criteria | week 24
Incidence of treatment-emergent Adverse Events | Up to week 36
Satisfaction scale (subjective satisfaction of patient and investigator with the treatment on a 5 Point likert scale) | week 1, week 12, week 24, week 36
  Subjective satisfaction on a scale from 1 (very satisfied) to 5 (very unsatisfied)

CONTACTS AND LOCATIONS:
Overall Officials: Dr. med. Eichhorn, Principal Investigator — Praxiszentrum Elisengalerie
Locations (1):
- Praxiszentrum Elisengalerie, Aachen, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lynen NA, Eichhorn C, Portelange N, Chausson M, Weyenberg W. Long-Term Efficacy Following Intra-articular Injection of Carboxymethyl-chitosan, a New Product Class for Knee Osteoarthritis: Results from an Observational Study in Germany. Rheumatol Ther. 2024 Jun;11(3):649-662. doi: 10.1007/s40744-024-00661-6. Epub 2024 Mar 18. PMID 38498142